CLINICAL TRIAL: NCT01187160
Title: A Pilot Study Assessing Surgical Exposure During Transoral Robotic Surgery (TORS) for Sleep Apnea Using the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA)
Brief Title: Transoral Robotic Surgery (TORS) for Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 809623
Record Dates: First submitted 2010-02-19; First posted 2010-08-23 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transoral robotic surgery (TORS) (Experimental): da Vinci® Robotic Surgical System
  Interventions: Procedure: Transoral robotic surgery (TORS)

INTERVENTIONS:
Procedure: Transoral robotic surgery (TORS) — The da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) is a manual image-guided surgery system that is computer enhanced rather than computer guided robotic surgery in which the surgeon programs the computer to do the surgery and the robot does the surgery (also known as a milling device). Use of the da Vinci® Robotic Surgical System in the aforementioned configuration in fact facilitates an exact translation of the surgeons hand and finger movements at the console to precise and tremor-free movements of the arms and instruments.
  Other Names: da Vinci® Robotic Surgical System

SUMMARY:
The purpose of this study is to assess if the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) allows for "adequate exposure" for transoral resection of hypertrophic lingual tonsils in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Visit 1 - Outpatient Clinical Setting. The patient will be evaluated prior to treatment in the outpatient clinical setting in a way which is consistent for routine workup prior to any surgery of the tongue base for sleep apnea. This will include sleep nasendoscopy (see below), and if it is predicted pre-treatment that the transoral robotic approach may be appropriate then the patient will be given the option of participating in the study. This will include a review of the patient's pre-operative sleep study and a nasopharyngolaryngoscopic exam to assess for lingual tonsillar hypertrophy. A pre-operative MRI will be obtained to provide quantitative measurement of the patient's tongue base hypertrophy.

Visit 2 - Sleep Nasendoscopy. The patient will undergo sleep nasendoscopy as outlined below, in order to assess the involvement of the tongue base in the patient's sleep disordered breathing. This is a routine diagnostic procedure. Patients are pharmacologically induced into a light phase of sleep and the upper airway is visualized directly with a nasopharyngolaryngoscope. Anesthetic management will be performed in standard fashion, using propofol titrated to an endpoint of moderate sedation, as is typically done for procedural sedation in esophagogastroduodenoscopy. Administration will be logged to permit analysis of dosing requirements. Respiratory pattern will be monitored noninvasively and logged to permit correlation of obstruction to propofol administration.

Visit 3 - Intraoperative Setting. The patient will undergo an evaluation for "adequate exposure" for transoral robotic surgery and if "adequate exposure" is achieved then they will undergo transoral robotic surgery for lingual tonsillar hypertrophy to treat obstructive sleep apnea.

Visit 4 - Postoperative Setting. This will be in the inpatient and/or outpatient setting within three weeks of surgical procedure. The patient will undergo routine postoperative clinical evaluation.

Visit 5 - Postoperative Testing. The patient will undergo a follow-up sleep study to determine efficacy of the surgical procedure at three months post-operatively, the standard interval used to determine the outcome of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 or older at time of treatment.
* Patient must present with indications for surgical management of the tongue base to treat obstructive sleep apnea.
* Written informed consent and/or consent waiver by IRB.

Exclusion Criteria:

* Pre-operative exclusion criteria:
* Unexplained fever and/or untreated, active infection.
* Patient pregnancy.
* Previous head and neck surgery precluding transoral/robotic procedures.
* The presence of medical conditions contraindicating general anesthesia or transoral surgical approaches.
* Intra-operative exclusion criteria (It is recognized that sometimes patients cannot be excluded from study participation until prepared in the surgical suite such that their anatomy is exposed and available for medical analysis. The following situations represent instances whereby patients would be excluded from this study based upon anatomical findings not evident in the pre-operative setting):
* Inability to adequately visualize anatomy to perform the diagnostic or therapeutic surgical approach transorally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To assess if the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) allows for "adequate exposure" for transoral resection of hypertrophic lingual tonsils in patients with obstructive sleep apnea. | 1 year

SECONDARY OUTCOMES:
To assess ability to perform the transoral diagnostic removal of hypertrophic lingual tonsils using the robotic system for transoral resection of the tongue base in patients with obstructive sleep apnea. | 1 year
To assess operative time to perform the transoral diagnostic removal of hypertrophic lingual tonsils using the robotic system for transoral resection of the tongue base in patients with obstructive sleep apnea. | 1 year
To assess blood loss during the transoral diagnostic removal of hypertrophic lingual tonsils using the robotic system for transoral resection of the tongue base in patients with obstructive sleep apnea. | 1 year
To assess complications of the transoral diagnostic removal of hypertrophic lingual tonsils using the robotic system for transoral resection of the tongue base in patients with obstructive sleep apnea. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erica Thaler, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States